CLINICAL TRIAL: NCT02588430
Title: Post-Market Clinical Follow-up Study for Partial Vision Restoration Using the Subretinal Implant RETINA IMPLANT Alpha AMS
Brief Title: PMCF Study for Partial Vision Restoration Using the Subretinal Implant RETINA IMPLANT Alpha AMS
Status: Withdrawn | Type: Observational
Why Stopped: Manufacturer of the investigational device has ceased all business activities
Sponsor: Retina Implant AG (Industry)
Responsible Party: Sponsor
Other Study IDs: RI-PMCF1-EU
Record Dates: First submitted 2014-09-30; First posted 2015-10-27 (Estimated); Last update posted 2019-04-19 (Actual); Status verified 2019-04

CONDITIONS: Retinitis Pigmentosa
MeSH Terms: conditions — Retinitis Pigmentosa

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Years
Oversight: Data Monitoring Committee: No

SUMMARY:
This study is a post-market clinical follow-up (PMCF) study to monitor the safety, lifetime and efficacy of patients using the CE-certified RETINA IMPLANT Alpha AMS.

DETAILED DESCRIPTION:
This study is a post-market clinical follow-up (PMCF) study to monitor the safety, lifetime and efficacy of patients using the CE-certified RETINA IMPLANT Alpha AMS. For Germany, it is under the exceptions mentioned in §23b MPG (Medizinproduktegesetz, German Medical Device Law). Its purpose is to collect data that is created during the regular therapy with the implant. No additional examinations are performed, except a patient questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Patients who received a RETINA IMPLANT Alpha AMS.
* Patients willing and able to give written informed consent.

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who received a Retina Implant Alpha at the study site. Patients who are fulfilling specific criteria to receive a RETINA IMPLANT Alpha AMS.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2019-03 (Estimated); Primary Completion 2029-12 (Estimated); Study Completion 2030-06 (Estimated)

PRIMARY OUTCOMES:
Time to device failure | 6 Years
  Recording of device failures
Number, nature and severity of challenges or complications during surgical procedures | 6 Years
  Recording of adverse events
Number, nature and severity of device-related adverse events and incidents until device failure or explantation | 6 Years
  Recording of adverse events

SECONDARY OUTCOMES:
1. Functional Vision Test | 6 Years
  Eye-hand coordination: a cup should be placed in the middle of a plate
2. Functional Vision Test | 6 Years
  Activity of daily living - Table test: 4 white items of big plate, small plate, bowl, cup and cutlery are placed on a black table cloth and should be identified and touched
3. Functional Vision Test | 6 Years
  Activity of daily living - Clothes sorting: socks in white, grey and black should be sorted
4. Functional Vision Tests | 6 Years
  Assessment of grating acuity: cards with grid patterns of different widths are presented and should be described
Visual related quality of life (Patient reported outcome) | 6 Years
  Impact of Vision Impairment - Very Low Vision Questionnaire (IVI-VLV) (Finger et al., 2014) is asking for vision-related quality of life by rating impact of eyesight on various tasks, referring to the last month

CONTACTS AND LOCATIONS:
Overall Officials: Florian Gekeler, Prof Dr med, Principal Investigator — Katharinenhospital Stuttgart
Locations (1):
- Katharinenhospital Stuttgart, Stuttgart, Germany

REFERENCES:
- [Background] Stingl K, Bartz-Schmidt KU, Besch D, Braun A, Bruckmann A, Gekeler F, Greppmaier U, Hipp S, Hortdorfer G, Kernstock C, Koitschev A, Kusnyerik A, Sachs H, Schatz A, Stingl KT, Peters T, Wilhelm B, Zrenner E. Artificial vision with wirelessly powered subretinal electronic implant alpha-IMS. Proc Biol Sci. 2013 Feb 20;280(1757):20130077. doi: 10.1098/rspb.2013.0077. Print 2013 Apr 22. PMID 23427175
- [Background] Koitschev A, Stingl K, Bartz-Schmidt KU, Braun A, Gekeler F, Greppmaier U, Sachs H, Peters T, Wilhelm B, Zrenner E, Besch D. Extraocular Surgical Approach for Placement of Subretinal Implants in Blind Patients: Lessons from Cochlear-Implants. J Ophthalmol. 2015;2015:842518. doi: 10.1155/2015/842518. Epub 2015 Dec 10. PMID 26783453
- [Background] Stingl K, Bartz-Schmidt KU, Besch D, Chee CK, Cottriall CL, Gekeler F, Groppe M, Jackson TL, MacLaren RE, Koitschev A, Kusnyerik A, Neffendorf J, Nemeth J, Naeem MA, Peters T, Ramsden JD, Sachs H, Simpson A, Singh MS, Wilhelm B, Wong D, Zrenner E. Subretinal Visual Implant Alpha IMS--Clinical trial interim report. Vision Res. 2015 Jun;111(Pt B):149-60. doi: 10.1016/j.visres.2015.03.001. Epub 2015 Mar 23. PMID 25812924